CLINICAL TRIAL: NCT07068321
Title: Effects Of Godelieve Denis-Struf (GDS) Method Along With Cognitive Behavioral Therapy Through Smartphone Health App For Patients With Chronic Lumbosacral Discogenic Pain.
Brief Title: Effects Of GDS Method Along With CBTThrough Smartphone Health App For Patients With Chronic LDP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PhDRSW/Batch-Fall23/2221
Record Dates: First submitted 2025-07-07; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Lumbosacral Disc Syndrome
MeSH Terms: interventions — Control Groups; Transcutaneous Electric Nerve Stimulation; Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (transcutaneous electrical nerve stimulation) (Experimental)
  Interventions: Combination Product: Control Group (transcutaneous electrical nerve stimulation)
- Godelieve Denis-Struf (Active Comparator)
  Interventions: Combination Product: Godelieve Denis-Struf
- Godelieve Denis-Struf + Cognitive Behavioral Therapy (Active Comparator)
  Interventions: Combination Product: Godelieve Denis-Struf + Cognitive Behavioral Therapy

INTERVENTIONS:
Combination Product: Control Group (transcutaneous electrical nerve stimulation) — Control Group will consist of 20 sessions of 30 min, applied twice per week over a period of 3 months including transcutaneous electrical nerve stimulation, and standardized exercises for LBP through smart phone application.
  Arms: Control Group (transcutaneous electrical nerve stimulation)
Combination Product: Godelieve Denis-Struf — Experimental Group will receive 20 sessions of 30 min applied twice per week over a period of 3 months of GDS treatment through smart phone application.
  Arms: Godelieve Denis-Struf
Combination Product: Godelieve Denis-Struf + Cognitive Behavioral Therapy — Experimental Group 2 will receive 20 sessions of 45 min applied twice per week over a period of 3 months of GDS along CBT treatment through smart phone application.
  Arms: Godelieve Denis-Struf + Cognitive Behavioral Therapy

SUMMARY:
Chronic lumbosacral discogenic pain is a common and debilitating condition that significantly affects the quality of life of patients. Traditional treatments often focus on pain management, but a holistic approach combining physical exercises and psychological therapy can offer more sustainable relief.

DETAILED DESCRIPTION:
The Godelieve Denis-Struf (GDS) method has been shown to improve posture, mobility, and muscular imbalances in patients with musculoskeletal pain. Cognitive Behavioral Therapy (CBT) is another effective intervention that addresses the psychological factors contributing to chronic pain. With the rise of digital health solutions, smartphone applications have emerged as convenient tools to deliver these therapeutic methods. This study explores the combined effects of GDS exercises and CBT via a smartphone health app for individuals suffering from chronic lumbosacral discogenic pain.

ELIGIBILITY:
Inclusion Criteria:

* Age of 40 to 65 years
* Diagnosed chronic lumbosacral discogenic pain by a physician or neuro-physician.
* No surgical history of lumbosacral area

Exclusion Criteria:

* Pregnancy
* Diagnosis of cancer
* Fibromyalgia or inflammatory disease (eg, rheumatoid arthritis or spondylitis)
* Surgical cases of lumbosacral area
* comorbidity like uncontrolled diabetes and blood pressure

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2025-04-17 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
The Oswestry Disability Index (ODI) | 18 Months
  The Oswestry Disability Index (ODI) is a questionnaire used to assess the impact of low back pain on a person's daily life. It consists of 10 sections, each with six statements, and patients select the statement that best describes their situation. Each section is scored from 0 to 5, with 0 indicating no disability and 5 indicating the worst imaginable disability. The total score is then calculated and can be expressed as a percentage, with a higher score indicating greater disability
SF-36 (Short Form 36) | 18 Months
  The SF-36 (Short Form 36) is a questionnaire used to assess health-related quality of life, encompassing both physical and mental well-being. It consists of 36 items that evaluate eight health domains: physical functioning, role limitations due to physical health, bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional problems, and mental health. Scores for each domain range from 0 to 100, with higher scores indicating better health

CONTACTS AND LOCATIONS:
Locations (1):
- Rehabilitation Centers in Punjab, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No